CLINICAL TRIAL: NCT04115865
Title: Assessment of Post-operative Sore Throat After Scheduled General Anesthesia
Acronym: POST
Status: Withdrawn | Type: Observational
Why Stopped: refusal ethics comity
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_96; 2019-A02077-50 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Sore Throat; Intubation;Difficult
MeSH Terms: conditions — Pharyngitis | interventions — Laryngeal Masks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endotracheal sonde or laryngeal mask — Healthy subjects ; requiring general anesthesia with endotracheal or endobuccal device

SUMMARY:
Precise description of the technique for intubation or laryngeal mask placement during general anesthesia Research on factors that can influence sore throat due to the placement of an endobuccal or endotracheal device during general anesthesia

ELIGIBILITY:
Inclusion Criteria:

- General Anesthesia required Endotracheal or endobuccal device

Exclusion Criteria:

* Tracheotomy per or post surgery
* Patient with pre-operative pharyngeal irritation.
* Patient with a prior respiratory tract infection.
* Surgery of the laryngeal or tracheal vein, old or new
* Surgery scheduled less than 24 hours ago.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient to be operated on in the Department of Surgical Specialties, Neurosurgery, Orthopaedics and Pediatric Surgery at the University Hospital of Lille
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of sore throat | Within 24 hours of surgery

SECONDARY OUTCOMES:
Severity of sore throat, | At exit of the post-interventional monitoring room, at 24 hours of surgery or exit of hospital
type of sore throat risk factor | At exit of the post-interventional monitoring room, at 24 hours of surgery or exit of hospital
  (technique of intubation, analgesic treatment for surgery…)

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Jozefowicz, MD, Principal Investigator — University Hospital, Lille